CLINICAL TRIAL: NCT06406465
Title: A UGT1A1 Genotype-Directed Study of Belinostat Pharmacokinetics and Toxicity
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10001601; 001601-C
Record Dates: First submitted 2024-05-08; First posted 2024-05-09 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-15

CONDITIONS: Carcinoma, Neuroendocrine; Tumor, Neuroendocrine; Tumors, Neuroendocrine; Neuroendocrine; Carcinoma; Small Cell; Receptors
Keywords: High-grade carcinomas; Resemble small cell carcinoma; Large cell NEC; Histone Deacetylase; Genotypes; Neuroendocrine malignancies
MeSH Terms: conditions — Carcinoma, Neuroendocrine; Neuroendocrine Tumors | interventions — belinostat; Cisplatin; Etoposide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Belinostat at 400 mg/m^2/day plus Cisplatin plus Etoposide
  Interventions: Drug: Belinostat; Drug: Cisplatin; Drug: Etoposide
- Arm 2 (Experimental): Belinostat at 600 mg/m^2/day plus Cisplatin plus Etoposide
  Interventions: Drug: Belinostat; Drug: Cisplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Belinostat — 400mg/m^2/24h or 600 mg/m^2/24h IV over (48h continuous infusion) on days 1, 2 and 3 based on UGT1A1 status
Drug: Cisplatin — 60 mg/m^2 IV over 60 minutes on day 2
Drug: Etoposide — 80 mg/m^2 IV over 60 minutes on day 2 after infusion of cisplatin and again on days 3 and 4

SUMMARY:
Background:

High-grade neuroendocrine carcinomas (HGNEC) are cancers that develop in different parts of the body, including the digestive tract, genitals, neck, and head. One drug (belinostat), combined with 2 other drugs (etoposide and cisplatin), is approved to treat HGNEC. But some people may have a gene variant that affects how quickly their body gets rid of the drug; these people may do better with different dosages of belinostat.

Objective:

To test higher or lower doses of belinostat based on gene variants in people with HGNEC.

Eligibility:

People aged 18 years and older with HGNEC.

Design:

Participants will be screened. They will have a physical exam with blood tests. Some blood will be used for genetic testing. They will have imaging scans and a test of their heart function. Samples of tumor tissue may be collected.

All 3 study drugs (belinostat, etoposide, cisplatin) are given through a tube attached to a needle inserted into a vein. Treatment will be given in 21-day cycles.

For cycles 1 through 6: Participants will come to the clinic for the first 4 days. They will be given all 3 drugs. Imaging scans and other tests will be repeated. Each visit will last 4 to 8 hours.

After cycle 6: Participants may continue treatment with belinostat alone. They will come to the clinic for the first 3 days of each cycle. They may continue treatment for up to 5 years if the drug is helping them.

Participants will have a follow-up visit 30 days after their last dose of belinostat. Then they will receive follow-up visits by phone or email every 3 to 6 months.

DETAILED DESCRIPTION:
Background:

* Extrapulmonary High-Grade Neuroendocrine Neoplasms (HGNENs) are all high-grade neoplasms that may resemble small cell carcinoma or large cell Neuroendocrine Carcinomas (NEC) of the lung. Poorly differentiated NECs are often associated with a rapidly progressive disease and a proliferative rate (Ki67%) >20%.
* As a general rule, poorly differentiated NECs are treated with platinum-based regimens according to small cell carcinoma guidelines.
* This protocol will study a continuous infusion of the histone deacetylase (HDAC) inhibitor belinostat in combination with cisplatin and etoposide for patients with advanced neuroendocrine neoplasms.

Objective:

-To determine if pharmacogenomic intervention can normalize the area under the curve (AUC) at cycle 6 between UGT1A1*28 and UGT1A1*60 genotypes) of belinostat administered as a continuous 48 h infusion in combination with cisplatin and etoposide in participants with neuroendocrine malignancies based on UGT1A1*28 and UGT1A1*60 genotypes.

Eligibility:

* The protocol will be open to participants with Extrapulmonary High-Grade Neuroendocrine Neoplasms (HGNENs)
* Participants will be recruited based on genotype, with n=9 carrying UGT1A1*1/*1 or UGT1A1*1/*28 and n=30 carrying any other combination of variant alleles at UGT1A1*28 or UGT1A1*60.
* Age >=18 years
* ECOG Performance Status 0-2

Design:

* Parallel design in which the starting dose of belinostat is administered as a 48-hour continuous infusion at two possible doses based on genotype: 1) 400mg/m^2/day for UGT1A1*28/*28 or at least one UGT1A1*60 allele UGT1A1*28 and UGT1A1*60 genotypes or 2) 600 mg/m^2/day for wild-type participants and those carrying UGT1A1*1/*28 in the absence of other variant alleles.
* To define pharmacokinetics, toxicities of belinostat provided to participants who carry the above genotype groups.
* All participants will also receive cisplatin at 60 mg/m^2 IV on day 2, and etoposide at 80 mg/m^2 IV daily x3 on days 2 - 4.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Participants must have histologically confirmed diagnosis of Extrapulmonary High-Grade Neuroendocrine Neoplasms (HGNENs) for which there is no known standard therapy capable of extending life expectancy.
2. Age >= 18 years.
3. Participants with neuroendocrine prostate cancer may continue ongoing LHRH agonist therapy.
4. Participants with bone metastases or hypercalcemia who began intravenous bisphosphonate treatment prior to study entry may continue this treatment while on study.
5. Evaluable (measurable or non-measurable) disease, per RECIST 1.1.
6. ECOG performance status <=2 at screening
7. Participants must have adequate organ and marrow function as defined below:

   * Leukocytes >=3,000/mcL
   * Hemoglobin >= 10 g/dL
   * Absolute neutrophil count (ANC) >=1,500/mcL
   * Platelets >=100,000/mcL
   * Aspartate aminotransferase (AST) or serum glutamic-oxaloacetic transaminase (SGOT) / Alanine aminotransferase (ALT) or serum glutamic-pyruvic transaminase (SGPT): <=3 X institutional upper limit of normal
   * Total bilirubin <= 1.5 x institutional upper limit of normal (ULN).

   NOTE: In participants with Gilbert s syndrome, a total bilirubin <= 3.0 X ULN is allowed
   * Serum Creatinine <= 1.5 X institutional ULN OR
   * An estimated Creatinine clearance (CrCL) >=60 mL/min/1.73 m^2 based on the Cockcroft Gault equation
   * Prothrombin time (PT) / International normalized ratio (INR) and Partial thromboplastin time (PTT) <= 1 X institutional ULN
8. Hepatitis B virus (HBV)-infected participants can be enrolled if HBV DNA is undetectable. Hepatitis C virus (HCV)-infected participants can be enrolled if HCV RNA level is undetectable
9. Women of child-bearing potential (WOCBP) must agree to use effective contraception (hormonal, intrauterine device (IUD), tube ligation, a partner has had a previous vasectomy, abstinence) prior to study entry, during the study, and for 14 months for women after the last dose of the study drug(s). Men with partners of childbearing potential must agree to use effective contraception (abstinence, condoms, previous vasectomy) or request partners to use effective contraception (per above) during the study and for 11 months after the last dose of study therapy.
10. Breastfeeding participants must be willing to discontinue breastfeeding starting with prior to study entry, during the study, and for 3 months after the last dose of the study drug(s).
11. Willing to comply with study procedures and follow-up.
12. Participants must be able to understand and be willing to sign a written informed consent document.

EXCLUSION CRITERIA:

1. Participants with prior investigational drug, chemotherapy, immunotherapy or any prior radiotherapy (except for palliative bone directed therapy) within the past 14 days prior to the first drug administration. Additionally, FDA-approved hormonal therapy for the treatment or prevention of other malignancies (e.g., breast cancer, prostate cancer) may be continued where in the opinion of the investigator stopping such therapies may increase the risk of disease progression. Potential drug-drug interactions with the hormonal agent will be assessed by the investigator prior to enrollment.
2. History of allergic reactions attributed to compounds of similar chemical or biologic composition to belinostat, cisplatin, etoposide or other agents used in study. Participants with a history of allergic reactions to medications containing polysorbate 80 will be evaluated on a case-by-case basis.
3. Participants with treated brain metastases are not eligible except if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression.
4. Participants who have not recovered (CTCAE <= grade 1) from non heme adverse events due to prior treatments, except for alopecia, or stable grade 2 tinnitus (not interfering with ADL's) or baseline hearing loss by audiometry or stable grade 2 sensory neuropathy (moderate symptoms; limiting instrumental ADL) without pain or motor component, and not interfering with ADL's.
5. Participants taking strong UGT1A1 inhibitors or CYP3A4 inhibitors or inducers must discontinue their use a minimum of 5 half-lives prior to starting treatment on this trial
6. Participants with platinum-refractory disease.
7. Participants who have had another histone deacetylase inhibitor (e.g., valproic acid, vorinostat) for at least 2 weeks prior to enrollment.
8. Participants who have had radiation to the pelvis or other bone marrow-bearing sites will be considered on a case-by-case basis and may be excluded if the bone marrow reserve is not considered adequate (>25% of bone marrow).
9. Pregnancy (confirmed with beta-Human chorionic gonadotropin (HCG) serum or urine pregnancy test performed in WOCBP at screening)
10. Significant cardiovascular disease (New York Heart Association Class III or IV cardiac disease), myocardial infarction within the past 6 months, unstable angina, unstable arrhythmia, or a need for anti-arrhythmic therapy (use of medication to control heart rate in participants with atrial fibrillation is allowed, if stable medication for at least last month prior to enrollment and medication not listed as causing Torsade de Points), or evidence of acute ischemia on ECG.
11. Baseline prolongation of QT/QTc interval, i.e., defined as an average QTc interval > 450 msec calculated using the Fridericia formula for QT correction; Long QT Syndrome; or the required use of concomitant medication that may cause Torsade de Pointes.
12. Participants with HIV infection if CD4 count <200 cells per cubic millimeter before treatment initiation
13. Uncontrolled intercurrent illness that would limit compliance with study requirements.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
To determine if pharmacogenomic intervention can normalize the area under the curve (AUC) at cycle 6 between UGT1A1*28 and UGT1A1*60 genotypes) of belinostat administered as a continuous 48 h infusion in combination with cisplatin and etoposide | Cycles 1-6 pre- and post- treatment with belinostat with all doses
  Identified as the PK parameter of interest.

SECONDARY OUTCOMES:
To determine efficacy with respect to objective response rate of belinostat administered as a continuous 48 h infusion in combination with cisplatin and etoposide | Every 9 weeks while on study therapy
  Objective response rate will be assessed by CT/MRI scans, calculated by Kaplan-Meier method, reporting the median values of each.
To determine the progression-free survival (PFS) and overall survival (OS) of belinostat administered as a continuous 48 h infusion in combination with cisplatin and etoposide | PFS will be assessed from on-study date until date of progression or death without progression. Overall survival (OS) will be calculated from the on-study date until date of death. Until 3 years after last participant enrolled.
  Progression free survival and overall survival calculated by Kaplan-Meier method, reporting the median values of each.
To assess duration of response of belinostat administered as a continuous 48 h infusion in combination with cisplatin and etoposide in platinum sensitive | Until progression or the response is declared to have ended , if the participants have a PR or CR. Until 3 years after last participant enrolled.
  Duration of response will be calculated by the Kaplan-Meier method, starting at date response was identified until progression or the response is declared to have ended, if the participants have a PR or CR.
To assess duration of response of belinostat maintenance | Every 9 weeks while on monotherapy. Total study therapy will not exceed 5 years.
  Duration of response will be calculated by the Kaplan-Meier method, starting at date response was identified until progression or the response is declared to have ended, if the participants have a PR or CR.

CONTACTS AND LOCATIONS:
Overall Officials: Jaydira Del Rivero, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review and/or will involve genomic data sharing. @@@@@@@@@@@@This study will comply with the NIH Genomic Data Sharing (GDS) Policy, which applies to all new and ongoing NIH IRP-funded research, as of January 25, 2015, that generates large-scale human or non-human genomic data, as well as the use of these data for subsequent research. Large-scale data include genome-wide association studies (GWAS), single nucleotide polymorphisms (SNP) arrays, and genome sequence, transcriptomic, epigenomic, and gene expression data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001601-C.html